CLINICAL TRIAL: NCT06652022
Title: Radiotherapy Combined with Systemic Therapy Versus Systemic Therapy for Oligometastatic Upper Tract Urothelial Carcinoma: a Prospective Randomised Controlled Trial
Brief Title: Radiotherapy Combined with Systemic Therapy Versus Systemic Therapy for Oligometastatic UTUCs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, LI xiaoying, Vice Director of the Department of Radiation Oncology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUXUS5.0
Record Dates: First submitted 2024-09-12; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Oligometastatic Disease; Ureter Cancer; Renal Pelvic Carcinoma
Keywords: Oligometastatic Disease; Upper tract urothelial carcinoma; systematic; radiotherapy; Randomized control trial
MeSH Terms: conditions — Ureteral Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systemic treatment group (Active Comparator): The choice of first-line treatment is based on the guidelines, and may include chemotherapy or immune checkpoint inhibitors, or a combination of therapies. For patients who can tolerate cisplatin, chemotherapy is given with the gemcitabine-cisplatin regimen, as follows: gemcitabine 1000mg/m2 d1,8; cisplatin 70 mg/m2, avoiding light, intravenous drip d2; 3 weeks for 1 cycle. For intolerant patients, the gemcitabine-carboplatin regimen is given as follows: gemcitabine 1000 mg/m2 d1,8, IV, carboplatin (4.5×[GFR+25]) mg, IV, d1; 3 weeks as 1 cycle. Immune checkpoint inhibitors and targeted agents may be administered if the patient does not tolerate chemotherapy; either in combination with chemotherapy or directly as first line.
  Interventions: Drug: Systematic drug treatment
- Systemic treatment combined with radiotherapy group (Experimental): For patients with oligometastases, the radiotherapy protocol adopts a full-coverage radiotherapy protocol for metastatic foci, which is used as early as possible during the 2 cycles of systemic treatment for the patients. For retroperitoneal lymph node metastases, the conventional segmental radiotherapy protocol is used, and for isolated metastatic foci, the SBRT radiotherapy is used as much as possible.
  PETCT was used to determine the location and number of metastatic foci before radiotherapy, and for some patients who could not undergo PETCT, chest, abdominal and pelvic CT, ultrasound of superficial lymph nodes, bone scanning and cranial MRI were used to define the scope of the patient's foci.
  Interventions: Radiation: Systematic therapy combined with radiotherapy

INTERVENTIONS:
Radiation: Systematic therapy combined with radiotherapy — Systematic medical therapy is same as the systematic treatment group. SBRT radiotherapy or conventional fractionated radiotherapy can be used according to the extent and size of the metastatic foci. SBRT radiotherapy is preferred, and a higher dose should be given as far as possible when the normal tissues permit, with a preferred single dose of ≥5Gy.
  Arms: Systemic treatment combined with radiotherapy group
Drug: Systematic drug treatment — The choice of first-line treatment is based on the guidelines, and may include chemotherapy or immune checkpoint inhibitors, or a combination of therapies. For patients who can tolerate cisplatin, chemotherapy is given with the gemcitabine-cisplatin regimen, as follows: gemcitabine 1000mg/m2 d1,8; cisplatin 70 mg/m2, avoiding light, intravenous drip d2; 3 weeks for 1 cycle. For intolerant patients, the gemcitabine-carboplatin regimen is given as follows: gemcitabine 1000 mg/m2 d1,8, IV, carboplatin (4.5×[GFR+25]) mg, IV, d1; 3 weeks as 1 cycle. Immune checkpoint inhibitors and targeted agents may be administered if the patient does not tolerate chemotherapy; either in combination with chemotherapy or directly as first line.
  Arms: Systemic treatment group

SUMMARY:
This study was a prospective, open-label, phase II randomised controlled clinical study, enrolling patients with primary oligometastatic uroepithelial carcinoma, oligometastasis was defined as ≤3 organs, and the number of metastatic lesions and size of metastases were not restricted to be able to satisfy the definition of full-coverage radiotherapy, with the exception of patients with brain metastases and more than 3 liver metastases.

If regional lymph node recurrence was present, all positive regional lymph nodes were collectively referred to as one lesion. Non-regional lymph node metastases were counted as the number of metastases by lymph node subregion.

Patients were divided into two groups according to whether they received radiotherapy or not: 1) systemic therapy group; 2) systemic therapy + radiotherapy group. Systemic drug therapy can be chosen from chemotherapy or immune checkpoint inhibitor therapy, or combination therapy.

DETAILED DESCRIPTION:
This study was a prospective, open-label, phase II randomised controlled clinical study, enrolling patients with primary oligometastatic uroepithelial carcinoma, oligometastasis was defined as ≤3 organs, and the number of metastatic lesions and size of metastases were not restricted to be able to satisfy the definition of full-coverage radiotherapy, with the exception of patients with brain metastases and more than 3 liver metastases.

If regional lymph node recurrence was present, all positive regional lymph nodes were collectively referred to as one lesion. Non-regional lymph node metastases were counted as the number of metastases by lymph node subregion.

Patients were divided into two groups according to whether they received radiotherapy or not: 1) systemic therapy group; 2) systemic therapy + radiotherapy group. Systemic drug therapy can be chosen from chemotherapy or immune checkpoint inhibitor therapy, or combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic uroepithelial cancer with histologically confirmed diagnosis (pathologically confirmed primary focus or one of the metastatic foci is sufficient) (metastasis after total cystectomy, metastasis after full-length nephroureteral resection, or metastatic uroepithelial cancer of the pelvic-ureteral bladder at the first diagnosis of inoperable metastatic uroepithelial cancer).
* Oligometastases were defined as ≤3 organs, and the number and size of metastatic lesions were not restricted to the extent that full-coverage radiotherapy could be met. If regional lymph node recurrence was present, all positive regional lymph nodes were collectively referred to as one lesion. Non-regional lymph node metastases are counted as metastases by lymph node subregion.
* Willing and able to provide written informed consent/assent for the trial; age ≥18 years on the date of signing the informed consent form and patient age ≤80 years.
* Expected survival time ≥ 6 months;
* Eastern Collaborative Oncology Group (ECOG) Physical Status (PS) score of 0 to 1;
* Normal major organ function, i.e., the following criteria are met: routine blood tests: a) Haemoglobin ≥ 90 g/L; b) Total bilirubin ≤ 2 x upper limit of normal (ULN); c) Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤ 2.5 x ULN in the absence of liver metastases, and ALT, AST and ALP ≤ 5 x ULN in the presence of liver metastases; d) Creatinine clearance (CrCl) ≥30 mL/min;

Exclusion Criteria:

* Pathological type non-urothelial carcinoma;
* Patients with brain metastases and >3 liver metastases; patients with spinal bone metastases at risk of spinal cord compression; patients with pericardial, pleural or abdominopelvic fluid;
* Patients who are intolerant to or have had a reduction in systemic therapy; patients with tumour progression assessed after 2 cycles of systemic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 1-year, 3-year and 5-year
  Tumour progression-free survival

SECONDARY OUTCOMES:
OS | 1-year, 3-year and 5-year
  Overall survival
Adverse effect | 1 month after the start of treatment until the end of treatment
  Adverse effect related to the therapies
ORR | 1-3 months after starting treatment
  Oncological response rate

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Departmeng of Urology, Peking University First Hospital, Beijing
  - Department of Radiotherapy Oncology, Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol